CLINICAL TRIAL: NCT04411693
Title: Prospective Randomized Comparative Trial for Combination Dexamethasone Implant With PRN Anti-VEGF Therapy to Anti-VEGF Therapy Alone in Treatment Resistant DME: Informing the Role for Imaging Biomarkers
Brief Title: Comparative Study of Dexamethasone Implant to Intravitreal Aflibercept in Subjects With Diabetic Macular Edema
Acronym: PRECISION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Justis Ehlers, The Norman C. and Donna L. Harbert Endowed Chair of Ophthalmic Research, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALLER1908JE
Record Dates: First submitted 2020-05-20; First posted 2020-06-02 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Intravitreal Dexamethasone Implant (Active Comparator): Subjects in this arm will be given intravitreal Dexamethasone implant injection at month 0. PRN intravitreal Dexamethasone implant injections will be given for persistent edema, if it has been 10 weeks or more since last implant injection. If it has been less than 10 weeks since last implant injection, subjects will receive PRN intravitreal Aflibercept for persistent edema.
  Interventions: Drug: Dexamethasone implant; Drug: Aflibercept
- Group B: Intravitreal Aflibercept (Active Comparator): Subjects in this arm will be given Intravitreal aflibercept at month 0. PRN intravitreal Aflibercept will be given at months 1-6 for persistent edema.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Dexamethasone implant — A sustained-release drug delivery system containing 0.7 mg of Dexamethasone. Implant is administered by intravitreal injection.
  Other Names: Ozurdex
  Arms: Group A: Intravitreal Dexamethasone Implant
Drug: Aflibercept — A single dose, 2mg, drug administered by intravitreal injection.
  Other Names: Eylea

SUMMARY:
This study is an interventional, prospective randomized study comparing the dexamethasone implant to intravitreal aflibercept. Subjects will have an initial single injection of aflibercept and will be randomized if diabetic macular edema persists. Each subject will be evaluated for 6 months following randomization. Thus, the study duration will be 12 months plus the recruitment period.

Subjects will be evaluated every month for safety, efficacy as measured by SDOCT and best corrected visual acuity (BCVA) using the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) protocol. In addition, ultra-widefield angiography will be performed at run-in visit, baseline, month 3, and month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent.
2. Men and women ≥ 18 years of age.
3. Foveal-involving retinal edema secondary to DME based on investigator review of SD-OCT.
4. Central subfield thickness on SDOCT of greater than or equal to 325 microns on Spectralis or 300 microns on Cirrus.
5. E-ETDRS best-corrected visual acuity of 20/400 or better in the study eye.
6. Willing, committed, and able to return for ALL clinic visits and complete all study related procedures.
7. Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) understand and willing to sign the informed consent form.

Exclusion Criteria:

1. Any prior or concomitant therapy with another investigational agent to treat DME in the study eye.
2. Prior panretinal photocoagulation in the study eye.
3. Prior intravitreal anti-VEGF therapy in the study eye.
4. Prior focal/grid laser photocoagulation in the study eye.
5. Prior history of intravitreal steroid therapy in the study eye.
6. Any history of severe allergy to fluorescein sodium (e.g., anaphylaxis, difficulty breathing) or other reason that the patient is unable to undergo fluorescein angiography (e.g., inability to get vascular access, unable to tolerate procedure). If allergy is mild and investigator believes can be pretreated with diphenhydramine to avoid allergic response, this is not an exclusion to enrollment.
7. Uncontrolled glaucoma at baseline evaluation (defined as intraocular pressure ≥25 mmHg despite treatment with anti-glaucoma medication) in the study eye and/or cup-to-disc ratio greater or equal to 0.8.
8. Active intraocular inflammation in either eye.
9. Active ocular or periocular infection in either eye.
10. Torn or ruptured posterior lens capsule in study eye. Laser capsulotomy is not a contraindication.
11. Prior systemic anti-VEGF therapy, investigational or FDA-approved, is only allowed up to 3 months prior to first dose, and will not be allowed during the study.
12. Significant vitreous hemorrhage obscuring view to the macula or the retinal periphery as determined by the investigator on clinical exam and ultra-widefield angiography, in study eye.
13. Presence of other causes of macular edema, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25 mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, choroidal neovascularization, age-related macular degeneration or multifocal choroiditis in the study eye. Epiretinal membranes are allowed.
14. Presence of macula-threatening traction retinal detachment in the study eye.
15. Prior vitrectomy in the study eye.
16. History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
17. Any history of macular hole of stage 2 and above in the study eye.
18. Any intraocular or periocular surgery within 3 months of Day 1 in the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as it's unlikely to interfere with the injection.
19. Prior trabeculectomy or other filtration surgery in the study eye.
20. Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.
21. Any history of uveitis in either eye.
22. Active scleritis or episcleritis in either eye.
23. Presence or history of scleromalacia in either eye.
24. Aphakia in the study eye.
25. Previous therapeutic radiation in the region of the study eye.
26. History of corneal transplant or corneal dystrophy in the study eye.
27. Significant media opacities, including cataract, in the study eye which might interfere with visual acuity, assessment of safety, or fundus photography.
28. Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the study period.
29. Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
30. Participation as a subject in any clinical study within the 12 weeks prior to Day 1.
31. Any systemic therapy with an investigational agent in the past 3 months prior to Day 1.
32. Any history of allergy to povidone iodine.
33. Pregnant or breast-feeding women
34. Women of childbearing potential* who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
The mean change in central subfield thickness | 6 months

SECONDARY OUTCOMES:
Number of injections | 6 months
Change in BCVA | 6 months
Change in leakage index | 6 months
Change in ischemic index | 6 months
Change in microaneurysm counts | 6 months
Change in ellipsoid zone integrity | 6 months
  Change in ellipsoid zone integrity as measured by EZ-RPE central subfield thickness
Change in intraretinal fluid volume | 6 months
Change in DRSS | 6 months
The incidence and severity of ocular and non-ocular adverse events and serious adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Consultants of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No